CLINICAL TRIAL: NCT02467608
Title: A Randomized, Double-Blind, Active Drug Controlled Study to Assess the Efficacy of HUEXC030 as Add-on Excipient to Eradicate Anti-Tuberculosis Drugs Induced Liver Injury in Subjects With Pulmonary Tuberculosis
Brief Title: Efficacy of HUEXC030 in Subjects With Pulmonary Tuberculosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Orient Pharma Co., Ltd. (Industry)
Collaborators: National Defense Medical Center, Taiwan (Other); National Research Program for Biopharmaceuticals, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NDMC HUEXC030-TB1
Record Dates: First submitted 2015-05-31; First posted 2015-06-10 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Pulmonary Tuberculosis
Keywords: HUEXC030; Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Isoniazid; NSC 366140

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isoniazid with HUEXC030 and RZE (Experimental): Subjects who are genotyped as high risk group will be receiving 2 months of intensive treatment comprised of 4 drugs (Isoniazid with HUEXC030 [H], rifampin [R], pyrazinamide [Z] and ethambutol [E]), followed by 4 months of continual chemotherapy consist of Isoniazid, Rifampin (2HRZE/4HR regimen). Subjects who are of low risk genotype will be removed from study after 8 weeks of study treatment, then return to conventional TB medication at least one follow-up visit at 4 weeks after the end of study treatment visit.
  Dosage is as below:
  Isoniazid with Isoniazid(H):300mg/600mg daily, rifampin [R]: 450~600mg daily, pyrazinamide [Z]; 1000~2000mg daily and ethambutol [E]: 800-1600mg daily)
  Interventions: Drug: Isoniazid with HUEXC030 and RZE
- Isoniazid (Other): Subjects who are genotyped as high risk group will be receiving 2 months of intensive treatment comprised of 4 drugs (Isoniazid [H], rifampin [R], pyrazinamide [Z] and ethambutol [E]), followed by 4 months of continual chemotherapy consist of Isoniazid, Rifampin (2HRZE/4HR regimen). Subjects who are of low risk genotype will be removed from study after 8 weeks of study treatment, then return to conventional TB medication at least one follow-up visit at 4 weeks after the end of study treatment visit.
  Dosage is as below:
  Isoniazid (H):300mg daily, rifampin [R]: 450~600mg daily, pyrazinamide [Z]; 1000~2000mg daily and ethambutol [E]: 800-1600mg daily)
  Interventions: Drug: HRZE

INTERVENTIONS:
Drug: Isoniazid with HUEXC030 and RZE — Subjects will receive oral study drug daily in accordance with the following regimen, that is, INH, RMP, PZA, and EMB for the first 2 months followed by INH, RMP and EMB (if medically indicated) daily for 4 additional months
  Other Names: INH with HUEXC030, RMP, PZA and EMB
  Arms: Isoniazid with HUEXC030 and RZE
Drug: HRZE — the same as experimental group,without the excipient of HUEXC030 only
  Other Names: INH, RMP, PZA and EMB
  Arms: Isoniazid

SUMMARY:
Assess the Efficacy of HUEXC030 as Add-on Excipient to Eradicate Anti-Tuberculosis Drugs Induced Hepatic Injury ( ATDH ) in Subjects with Pulmonary Tuberculosis

DETAILED DESCRIPTION:
The study drug is Isoniazid formulated with HUEXC030 as excipient for eradicating ATDH, whereas the reference control is Isoniazid formulated with inactive excipient. Subjects who fulfill all the entry criteria and have written informed consent will be enrolled to the study. Eligible subjects will be randomized in a 1:1 ratio to receive study drug or reference control drug. Subjects will be genotyped according to a selected panel of single nucleotide polymorphisms (SNPs) and categorized into high risk or low risk groups for occurring ATDH via a specific haplotype consists of CYP2E1 and NAT2 SNPs. Based on an extensive study result during 2007 to 2011,the estimated frequency for patients bearing high risk genotypes in Taiwanese population is around 25%. Approximately 352 subjects will be enrolled for genotype screening in order to recruit 88 high risk subjects for each of 44 subjects in the intervention and control arms.

Subjects who are stratified as high risk groups will be administered the test drug or reference control drugs oral daily for 6 months or until treatment completion, i.e. bacteriologically confirmed negative of active M. tuberculosis. Subjects who are of low risk genotype will be removed from study after 8 weeks of study treatment, then return to conventional TB medication under the care of their investigator for at least one follow-up visit at 4 weeks after the End of Study.

ELIGIBILITY:
Main inclusion criteria:

1. A definite case of pulmonary TB
2. Patient who is exposed to 3 or less doses of first-line anti-TB drug treatment for current disease.
3. Age ≥ 20 years
4. Have well documented baseline liver function tests that indicates patient's adequate liver function for enrollment to study.

   i. AST and ALT < 3x ULN ii. total serum bilirubin < 2.0 mg/dL

Main Exclusion Criteria:

1. Have alcoholic liver disease or habitual alcohol consumption > 30 g/day for more than one year
2. Previously diagnosed of:

   i. extra-pulmonary TB without concomitant lung invasion ii. HIV iii. liver malignancy iv. liver cirrhosis v. any other systemic diseases that may cause liver dysfunction
3. Documented history of serious allergic reaction or resistance to isoniazid, rifampicin, ethambutol, pyrazinamide, sugar alcohols or any structurally related compounds
4. Subjects who will be using the following therapies after TB treatment starts:

   i. antiretroviral agents ii. oral corticosteroids
5. Subjects are pregnant or lactating
6. Subjects with child-bearing potential who are not committed to take reliable contraception during the participation of the study and at least 4 weeks after the end of the study treatment
7. Subjects with any other serious disease considered by the investigator not in the condition to enter into the trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
ALT change from baseline to the 8 weeks of study treatment | 8 weeks
  The primary efficacy endpoint is the time-interval weighted area under the curve (AUC) of change from baseline in serum ALT, primarily in patients with high risk genotypes. The area under ALT change curve was estimated using the linear trapezoidal rule. The AUC was a measure of cumulative ALT differences from baseline to the 8 weeks of double-blind treatment period.

SECONDARY OUTCOMES:
Incidence of ATDH in high risk genotype subjects treated with investigational drugs | 8 weeks
  Primarily in patients with high risk genotypes, the lowering incidence of ATDH in subjects treated with anti-TB drugs in combination with HUEXC030 for 8 weeks.
Incidence of ATDH in high risk genotype subjects treated with investigational drugs | 26 weeks
  Primarily in patients with high risk genotypes, the lowering incidence of ATDH in subjects treated with anti-TB drugs in combination with HUEXC030 for 26 weeks or at treatment completion.
Percentage of patients cured by the end of treatment | 8 weeks
  At 8 weeks, the investigational product is not inferior in effectiveness of TB treatment to the control drug, primarily in patients with high risk genotypes.
Percentage of patients cured by the end of treatment | 26 weeks
  At 26 weeks or at treatment completion, the investigational product is not inferior in effectiveness of TB treatment to the control drug, primarily in patients with high risk genotypes.
The overall reduced incidence of ATDH in subjects treated with investigational drugs | 26 weeks
  Compared to control drugs, the overall reduced incidence of ATDH in all enrolled subjects treated with investigational drugs at study ends.
The lowering average level of liver function tests | 26 weeks
  Compared to control drugs, the lowering average level of liver function tests in all enrolled subjects treated with investigational drugs at study ends.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Pu Hu, PhD, Study Chair — National Defense Medical Center, Taiwan
Locations (18):
- Taiwan (18):
  - Changhua Christian Hospital, Changhua
  - Changhua Hosiptal Ministry of Health And Welfare, Changhua
  - Chang Gung Memorial Hospital, ChiaYi, Chiayi City
  - Chang Gung Memorial Hospital, Kaohsiung, Kaohsiung City
  - E-DA Hospital, I-Shou University, Kaohsiung City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital ,Linkou, Linkou District
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Buddhist Tzu Chi General Hospital, Taipei
  - Cheng Hsin General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei City Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Medical University-Shuang Ho Hospital, Taipei
  - Taipei Wanfang Hospital, Taipei